CLINICAL TRIAL: NCT02581761
Title: A Randomized Prospective Double Blind Study of Misoprostol Administration in Asymptomatic Patients With Pregnancies of Unknown Location
Brief Title: A Prospective Study of Misoprostol Administration in Asymptomatic Patients With Pregnancies of Unknown Location
Acronym: amalis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Isa Amal, DR, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: SHEBA-14-1327-IA-CTIL
Record Dates: First submitted 2015-08-27; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Pregnancies of Unknown Location (PUL)
Keywords: Hemodynamically stable women >18 years old; with abnormal plateauing serum βHCG
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cytotec treatment group (Experimental): patient with pregnancy of unkown location will receive cytotec 800 mcg per vaginal
  Interventions: Drug: CYTOTEC
- Placebo treatment group (Placebo Comparator): patient with pregnancy of unkown location will receive suppository which contain Whitepsol H-15 with no active material (Cytotec).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CYTOTEC — synthetic prostaglandin E1
  Other Names: Misoprostol
  Arms: Cytotec treatment group
Other: Placebo — no active material
  Other Names: Whitepsol H-15
  Arms: Placebo treatment group

SUMMARY:
A randomized prospective double blind study of misoprostol administration in asymptomatic patients with pregnancies of unknown location.

DETAILED DESCRIPTION:
A randomized prospective double blind study of misoprostol administration in asymptomatic patients with pregnancies of unknown location.

The management of asymptomatic patients with pregnancies of unknown location (PUL) remains a challenge. Determining the location of the pregnancy is the first priority in the evaluation of these women. Some of these asymptomatic women present with inappropriate raising beta-human chorionic gonadotropin (βHCG), while others have assurance of pregnancy duration (e.g. IVF pregnancies) with no sonographic evidence of intra or extra uterine pregnancy. Most of the PULs are failed intra-uterine pregnancies.

The main concern regarding PUL is the late diagnosis of an ectopic pregnancy (EP). Some studies report that between 5 and 42% of women seen for US assessment with a positive pregnancy test have a PUL and only 6-20% will subsequently diagnosed with EP (1). Other studies report that 94% of PUL will resolve spontaneously, and out of the 6% that did not spontaneously resolve 68.9 % were finally diagnosed with failed IUP and only 5.6% were diagnosed with EP (2).

Women with PUL should be evaluated in minimum time, but also with minimal invasiveness. Management that will resolve such pregnancies in a rapid manner will save time and money and possibly avoid unnecessary administration of MTX or surgical intervention.

Several protocols have been investigated in order to fasten the diagnosis of PUL. For example, obtaining serial β-HCG, the first one in the initial presentation, two days later and seven days later (3). Another protocol suggested endometrial sampling by D&C or aspiration of uterine continents with Karman cannula and checking the β-HCG after 24 hours (2).

Purpose: The aim of our study will be to prospectively assess the use of misoprostol in asymptomatic patients with pregnancies of unknown location(PUL).

The study group will contain hemodynamically stable women >18 years old with a PUL with abnormal plateauing serum β-HCG trend (increase<53%or decrease <15% in 2 days) < 1000 IU/l and a pelvic ultrasound unremarkable for an intrauterine pregnancy (IUP) or an ectopic pregnancy (EP).

Each participant will get Vaginal misoprostol 800 mcg or placebo. Main Outcome Measure(s): The primary outcome measure will be an uneventful decline of serum β-HCG to an undetectable level (<2 IU/l) by the initial intervention strategy. Secondary outcome measures will include additional treatment (e.g. methotrexate (MTX) administration or laparoscopy), side effects and serum β-HCG clearance time, features of the optimal candidates for treatment by cytotec.

ELIGIBILITY:
Inclusion Criteria:

* hemodynamically stable women >18 years old with a PUL with abnormal plateauing serum βHCG trend

Exclusion Criteria:

* Hemoglobin<10

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be an uneventful decline of serum β-HCG to an undetectable level (<2 IU/l) by the initial intervention strategy | two weeks for each patient